CLINICAL TRIAL: NCT02738853
Title: The Medtronic TAVR 2.0 US Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10233065DOC
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medtronic Transcatheter Aortic Valve 2.0 Replacement System (Experimental): Treatment of Aortic Stenosis by replacing native valve with the Medtronic Transcatheter Aortic Valve 2.0 System
  Interventions: Device: Medtronic Transcatheter Aortic Valve 2.0 Replacement System

INTERVENTIONS:
Device: Medtronic Transcatheter Aortic Valve 2.0 Replacement System — Treatment of severe symptomatic aortic stenosis in subjects who are considered at high through extreme risk for surgical aortic valve replacement.

SUMMARY:
The study objective is to evaluate safety and efficacy of the Medtronic TAVR (Transcatheter Aortic Valve Replacement) 2.0 system in patients with severe symptomatic aortic stenosis who are considered at high through extreme risk for surgical aortic valve replacement

DETAILED DESCRIPTION:
Prospective, single arm, multi-site study. Patients will be seen at pre and post procedure, discharge, 30 days, 6 months, 1 year, and annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis, defined as aortic valve area of <1.0 cm2 (or aortic valve area index of <0.6 cm2/m2) by the continuity equation, AND mean gradient >40 mmHg OR maximal aortic valve velocity >4.0 m/sec by resting echocardiogram
2. Society of Thoracic Surgeons(STS) score of ≥8 OR documented heart team agreement of ≥ high risk for aortic valve replacement due to frailty or co-morbidities
3. Symptoms of aortic stenosis AND New York Heart Association (NYHA) Functional Class II or greater
4. The subject and the treating physician agree that the subject will return for all required post procedure follow-up visits.

Exclusion Criteria:

1. Any condition considered a contraindication for placement of a bioprosthetic valve (eg, subject is indicated for mechanical prosthetic valve)
2. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre medicated:

   * aspirin or heparin (HIT/HITTS) and bivalirudin
   * ticlopidine and clopidogrel
   * nitinol (titanium or nickel)
   * contrast media
3. Blood dyscrasias as defined: leukopenia (WBC <1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states
4. Untreated clinically significant coronary artery disease requiring revascularization
5. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% by echocardiography, contrast ventriculography, or radionuclide ventriculography
6. End stage renal disease requiring chronic dialysis or creatinine clearance <20 cc/min.
7. Ongoing sepsis, including active endocarditis
8. Any percutaneous coronary or peripheral interventional procedure with a bare metal or drug eluting stent performed within 30 days prior to study procedure
9. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 10 weeks of Heart Team assessment
10. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support
11. Recent (within 6 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
12. Gastrointestinal (GI) bleeding that would preclude anticoagulation
13. Subject refuses a blood transfusion
14. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
15. Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions
16. Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams
17. Currently participating in an investigational drug or another device study (excluding registries)
18. Evidence of an acute myocardial infarction ≤30 days before the study procedure
19. Need for emergency surgery for any reason
20. Liver failure (Child-Pugh class C)
21. Subject is pregnant or breast feeding
22. Pre existing prosthetic heart valve in any position
23. Mixed aortic valve disease (aortic stenosis with severe aortic regurgitation)
24. Severe mitral regurgitation
25. Severe tricuspid regurgitation
26. Moderate or severe mitral stenosis
27. Hypertrophic obstructive cardiomyopathy
28. Echocardiographic or Multi-Slice Computed Tomography (MSCT) evidence of intracardiac mass, thrombus, or vegetation
29. Congenital bicuspid or unicuspid valve verified by echocardiography
30. Access vessel diameter <5.5 mm or <6.0 mm for patent left internal mammary artery (LIMA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Forrest, MD, Principal Investigator — Yale New Haven Hospital; Mathew Williams, MD, Principal Investigator — NYU Langone Medical Center
Locations (8):
- United States (8):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - The University of Kansas Hospital, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Morristown Memorial Hospital, Morristown, New Jersey
  - NYU / Langone Medical Center, New York, New York
  - New York-Presbyterian Hospital / Columbia University Medical Center, New York, New York
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wyler von Ballmoos MC, Reardon MJ, Williams MR, Mangi AA, Kleiman NS, Yakubov SJ, Watson D, Kodali S, George I, Tadros P, Zorn GL 3rd, Brown J, Kipperman R, Oh JK, Qiao H, Forrest JK. Three-Year Outcomes With a Contemporary Self-Expanding Transcatheter Valve From the Evolut PRO US Clinical Study. Cardiovasc Revasc Med. 2021 May;26:12-16. doi: 10.1016/j.carrev.2020.11.007. Epub 2020 Nov 10. PMID 33199247
- [Derived] Forrest JK, Mangi AA, Popma JJ, Khabbaz K, Reardon MJ, Kleiman NS, Yakubov SJ, Watson D, Kodali S, George I, Tadros P, Zorn GL 3rd, Brown J, Kipperman R, Saul S, Qiao H, Oh JK, Williams MR. Early Outcomes With the Evolut PRO Repositionable Self-Expanding Transcatheter Aortic Valve With Pericardial Wrap. JACC Cardiovasc Interv. 2018 Jan 22;11(2):160-168. doi: 10.1016/j.jcin.2017.10.014. PMID 29348010

RESULTS

PARTICIPANT FLOW:
Period: Enrollment
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 93
Completed | 60
Not Completed | 33
Not completed — Inclusion/Exclusion not met | 21
Not completed — Withdrawal by Subject | 3
Not completed — Subject treated with commercially available device | 6
Not completed — Study Enrollment Closed | 3
Period: Procedure
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 60
Completed | 59
Not Completed | 1
Not completed — Death | 1
Period: 1 Month
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 59
Completed | 57
Not Completed | 2
Not completed — Death | 2
Period: 6 Month
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 57
Completed | 51
Not Completed | 6
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2
Period: 1 Year
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 51
Completed | 44
Not Completed | 7
Not completed — Death | 6
Not completed — Withdrawal by Subject | 1
Period: 2 Year
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 44
Completed | 41
Not Completed | 3
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Period: 3 Year
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 41
Completed | 38
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Period: 4 Year
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 38
Completed | 29
Not Completed | 9
Not completed — Death | 9
Period: 5 Year
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Started | 29
Completed | 25
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Rate
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 1.7 [0.2 to 11.2]

2. Primary Outcome: Stroke (Disabling) Rate
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 1.7 [0.2 to 11.4]

3. Primary Outcome: The Percentage of Subjects With None or Trace Prosthetic Regurgitation on Echocardiogram
Time Frame: 30 days
Population: Only subjects with transthoracic echo (TTE) could be analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 58
percentage of participants | 72.4 [59.1 to 83.3]

4. Secondary Outcome: Event Rate of the VARC II Combined Safety Endpoint at 30 Days, Which Includes the Following Components:
Description: 1. All-cause mortality
     >
  2. All stroke (disabling and non-disabling)
     >
  3. Life-threatening bleeding
     >
  4. Acute kidney injury: stage 2 or 3 (including renal replacement therapy)
     >
  5. Coronary artery obstruction requiring intervention
     >
  6. Major vascular complication
     >
  7. Valve-related dysfunction requiring repeat procedure (BAV, TAVR, or SAVR)
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 15.0 [8.1 to 26.8]

5. Secondary Outcome: Percentage of Participants With Life Threatening or Disabling Bleeding
Description: Percentage of participants with life threatening or disabling bleeding - VARC-II definitions
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 11.7 [5.7 to 22.9]

6. Secondary Outcome: Percentage of Participants With Major Vascular Complication
Description: Percentage of participants with major vascular complication - VARC-II definition
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 10.0 [4.6 to 20.9]

7. Secondary Outcome: Percentage of Participants With Coronary Artery Obstruction
Description: Percentage of participants with coronary artery obstruction - VARC-II definitions
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 6.1]

8. Secondary Outcome: Percentage of Patient With Acute Kidney Injury- Stage 2 or 3
Description: Percentage of participants with Acute kidney injury - Stage 2 or 3 - VARC-II definitions
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 1.7 [0.2 to 11.2]

9. Secondary Outcome: Percentage of Participants With Valve-related Dysfunction Requiring Repeat Procedure
Description: Percentage of participants with valve-related dysfunction requiring repeat procedure - VARC-II definition
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 6.1]

10. Secondary Outcome: Device Success Rate (VARC II)
Time Frame: 24 hours to 7 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
percentage of participants | 80.8 [67.5 to 90.4]

11. Secondary Outcome: Hemodynamic Performance - Aortic Valve Area
Description: Aortic Valve Area (cm2) by transthoracic echocardiogram
Time Frame: 30 days
Population: Only subjects with TTE could be analyzed.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
cm2 | 2.0 (0.5)

12. Secondary Outcome: Hemodynamic Performance - Mean Gradient
Description: Mean gradient (mmHg) by transthoracic echocardiogram
Time Frame: 30 days
Population: Only subjects with TTE could be analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 60
mmHg | 6.4 (2.1)

13. Secondary Outcome: Hemodynamic Performance - Total Prosthetic Regurgitation Graded as None/Trace
Description: Total prosthetic regurgitation by transthoracic echocardiogram
Time Frame: 30 days
Population: Only subjects with TTE could be analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic Transcatheter Aortic Valve 2.0 Replacement System
Number analyzed (Participants) | 58
percentage of participants | 72.4

ADVERSE EVENTS:
Time Frame: All events 6 months, All Cause Mortality 60 months
Groups:
- TAVR 2.0: Participants implanted with the TAVR 2.0 system
Arm/Group | TAVR 2.0
All-Cause Mortality (participants affected / at risk) | 26/60
Serious Adverse Events (participants affected / at risk) | 39/60
Other Adverse Events (participants affected / at risk) | 38/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR 2.0 (N=60)
Anaemia (Blood and lymphatic system disorders) | 7 (8)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Atrioventricular Block Complete (Cardiac disorders) | 8 (8)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Bundle Branch Block Left (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 3 (5)
Cardiac Perforation (Cardiac disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Device Embolisation (General disorders) | 1 (1)
Implant Site Haemorrhage (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Incision Site Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound Secretion (Injury, poisoning and procedural complications) | 2 (2)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 3 (3)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Mental Disorder (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 3 (3)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Graft (Surgical and medical procedures) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR 2.0 (N=60)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10)
Atrial Fibrillation (Cardiac disorders) | 6 (6)
Atrioventricular Block First Degree (Cardiac disorders) | 8 (8)
Bundle Branch Block Left (Cardiac disorders) | 21 (24)
Cardiac Failure Congestive (Cardiac disorders) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No